CLINICAL TRIAL: NCT02275520
Title: Comparison of NIO, BIG, EZ-IO, Jamshidi and Cook Intraosseous Devices in Adult Patients Under Resuscitation by Paramedics: a Randomized Crossover Manikin Trial.
Brief Title: Intraosseous Access
Acronym: NIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IO2014
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Intraosseus Access; Manikin; Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IO access (Other): Performed intraosseus access device during simulated cardiopulmonary resuscitation
  Interventions: Device: NIO Adult device; Device: Bone Iniection Gun; Device: EZ-IO; Device: Jamshidi Intraosseous Needle; Device: Cook Intraosseous Needle

INTERVENTIONS:
Device: NIO Adult device — IO access-1
  Other Names: NIO
Device: Bone Iniection Gun — IO access-2
  Other Names: BIG
Device: EZ-IO — IO access-3
Device: Jamshidi Intraosseous Needle — IO access-4
  Other Names: Jamshidi
Device: Cook Intraosseous Needle — IO access-5
  Other Names: Cook

SUMMARY:
The investigators will compare the success rates and time to successful IO access during simulated adult resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* paramedic
* more than 1 year experience in medicine

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
time to IO needle insertion | 1 day
  time from picking up a intraosseous access device, to successful IO needle insertion in the bone

SECONDARY OUTCOMES:
time to IO needle stabilization | 1 day
  time from picking up a intraosseus access device to correct fixation IO needle
time to intraosseuss infusion | 1 day
  begining with picking up a intraosseuss access device and ending with the IV line tubing was connected to the inseted IO needle
Ease of use | 1 day
  To access subjective opinion about the difficulty of the procedure, participants were asked to rate it on a visual analogue scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland